CLINICAL TRIAL: NCT07156019
Title: A Prospective, Single-center, Single-arm Phase II Study of Sintilimab in Combination With Surufatinib and Temozolomide in the Treatment of Advanced Neuroendocrine Carcinoma
Brief Title: Sintilimab in Combination With Surufatinib and Temozolomide in the Advanced Neuroendocrine Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24/371-4651
Record Dates: First submitted 2024-12-21; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Neuroendocrine Carcinomas (NEC)
Keywords: Surufatinib; Temozolomide; Sintilimab; Neuroendocrine carcinomas; Prospective observational study
MeSH Terms: conditions — Carcinoma, Neuroendocrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Surufatinib + Surufatinib + Sintilimab (Experimental): After fully informed and signed informed consent, subjects will receive Sintilimab (200mg each fixed dose, once every 21 days) combined with Temozolomide (body surface area（BSA）≤1.7m2; BSA >1.7m2 was administered with 300mg, once daily, d1-d5, and with Surufatinib (250mg, once daily, continuous administration). A treatment cycle of 21 days until disease progression, death, toxicity intolerance or withdrawal of informed consent, with a maximum treatment period of 24 months.
  Interventions: Drug: Sintilimab+Temozolomide+Surufatinib

INTERVENTIONS:
Drug: Sintilimab+Temozolomide+Surufatinib — After fully informed and signed informed consent, subjects will receive Sintilimab (200mg each fixed dose, once every 21 days) combined with Temozolomide (BSA≤1.7m2; BSA > 1.7m2 was administered with 300mg, QD, d1-d5, and with Surufatinib (250mg, QD, continuous administration). A treatment cycle of 21 days until disease progression, death, toxicity intolerance or withdrawal of informed consent, with a maximum treatment period of 24 months.

SUMMARY:
This study will evaluate the efficacy, safety and tolerability of Surufatinib + Temozolomide + Sintilimab in subjects. A treatment cycle of 21 days until disease progression, death, toxicity intolerance or withdrawal of informed consent, with a maximum treatment period of 24 months. Efficacy evaluation was performed at the end of every 2 treatment cycles. After termination of study treatment, participants will be followed up for safety and survival (survival follow-up every 90 days).

DETAILED DESCRIPTION:
This study will evaluate the efficacy, safety and tolerability of Surufatinib + Temozolomide + Sintilimab in subjects. After fully informed and signed informed consent, subjects will receive Sintilimab (200mg each fixed dose, once every 21 days) combined with Temozolomide (body surface area（BSA）≤1.7m2; BSA >1.7m2 was administered with 300mg, once daily, d1-d5, and with Surufatinib (250mg, once daily, continuous administration). A treatment cycle of 21 days until disease progression, death, toxicity intolerance or withdrawal of informed consent, with a maximum treatment period of 24 months. Efficacy evaluation was performed at the end of every 2 treatment cycles. For subjects whose disease progression was evaluated for the first time according to Response Evaluation Criteria in Solid Tumors, version 1.1（RECIST v1.1）, the investigator determined that the subjects were clinically stable and still had clinical benefit, the subjects could continue to receive treatment, and the disease progression was confirmed according to Immune Response Evaluation Criteria in Solid Tumors（iRECIST） criteria 4-6 weeks later. After termination of study treatment, participants will be followed up for safety and survival (survival follow-up every 90 days).

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily joined the study, signed the informed consent, and the compliance was good;
2. Locally advanced unresectable or metastatic neuroendocrine carcinoma confirmed by histopathology or cytology (excluding small cell lung cancer);
3. Disease progression or toxicity intolerance after previous first-line and above treatment;
4. At least one measurable lesion according to RECIST v1.1;
5. Eastern Cooperative Oncology Group Performance Status（ECOG PS） score is 0-1;
6. Age ≥18 and ≤75 years old;
7. Can provide tumor specimens for biomarker detection；
8. Major organ and bone marrow function levels meet the following requirements within 7 days prior to treatment:

   ① Blood routine: Absolute neutrophil count (ANC) ≥1.5×10^9/L; Platelet count (PLT) ≥90×10^9/L; Hemoglobin (Hb) ≥9.0 g/dL; Have not received transfusions of blood products (including erythrocyte and platelet products, etc.) and have not used supportive therapy of growth factors (including colony-stimulating factor, interleukin and erythropoietin, etc.) within 2 weeks before the examination;

   ② Liver function: serum total bilirubin (TBIL) ≤1.5× upper limit of normal value (ULN); alanine Aminotransferase（ALT） and aspartate aminotransferase (AST) in subjects without liver metastasis ≤3.0×ULN, and ALT and AST in subjects with liver metastasis ≤5.0×ULN;

   ③ Renal function: serum creatinine (Cr) ≤1.5×ULN;

   ④ Coagulation function: International standardized ratio (INR) ≤1.5×ULN, and activated partial thromboplastin time (APTT) ≤1.5×ULN;

   ⑤ Urine routine results showed that urine protein <2+; For patients with urine protein ≥2+ in routine urine testing at baseline, a 24-hour urine protein quantity of <1g is required;
9. Expected survival time ≥3 months;
10. Women of reproductive age should agree to use contraceptives (such as Iuds, contraceptives, or condoms) during the study period and for 6 months after the study ends; Have a negative serum or urine pregnancy test within 7 days prior to study enrollment and must be a non-lactating patient; Men should consent to patients who must use contraception during the study period and for 6 months after the end of the study period.

Exclusion Criteria:

1. Previous exposure to any anti-PD-1 /PD-L1/PD-L2/CTLA-4 antibody, VEGF/VEGFR targeting drugs;
2. Previous treatment with temozolomide;
3. Received chemotherapy, targeted therapy, Chinese herbal medicine with anti-tumor indications, or immunomodulatory drugs within 4 weeks prior to enrollment, or remained within 5 half-lives of such drugs;
4. Known to be allergic to any monoclonal antibody, temozolomide preparations, and solfantinib preparations;
5. Use of immunosuppressive drugs within 4 weeks prior to initial administration, excluding nasal, inhalation, or other routes of local corticosteroids or physiological doses of systemic corticosteroids;
6. There was toxicity caused by previous anti-tumor therapy that did not recover to NCI CTCAE5.0 version ≤ Grade 1 before the first administration;
7. History of other primary malignancies, except the following: non-melanoma skin cancer or malignant lentigo with adequate treatment and no evidence of disease recurrence, carcinoma in situ with adequate treatment and no evidence of disease recurrence;
8. Patients with metastatic central nervous system or cancerous meningitis with clinical symptoms;
9. Hepatic encephalopathy, hepatorenal syndrome or Child-Pugh grade B or more severe cirrhosis;
10. Inability to swallow, intestinal obstruction, or other factors affecting the administration and absorption of the drug;
11. Have serious heart disease or discomfort;
12. The patient has any active autoimmune disease or a history of autoimmune disease within 2 years;
13. Pregnant or nursing female patients;
14. A history of immunodeficiency, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
15. Had undergone major surgery within 4 weeks prior to enrollment or expected to require major surgery during the study treatment;
16. Concurrent participation in another interventional clinical study, unless participating in an observational (non-interventional) clinical study or in the follow-up phase of an interventional study;
17. Has a serious concomitant disease or other comorbidities that interfere with planned treatment;
18. Any other circumstances deemed inappropriate for participation in this study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | From enrollment to the end of treatment at 1 year
  Objective response rates assessed according to RECIST v1.1 criteria. It defines as the proportion of patients who achieve either a Complete Response (CR) or Partial Response (PR) of total evaluable patients.

SECONDARY OUTCOMES:
Progression-free survival | From enrollment to the end of treatment at 1 year
  Time from randomization/treatment initiation to disease progression (PD), or death from any cause (whichever occurs first).
Disease control rates | From enrollment to the end of treatment at 1 year
  The proportion of patients who achieve Complete Response (CR), Partial Response (PR), or Stable Disease (SD).
Overall survival | From enrollment to the end of treatment at 1 year
  The time from randomization/treatment initiation to death from any cause.
Incidence of Treatment-Emergent Adverse Events | From enrollment to the end of treatment at 1 year
  Incidence and severity of adverse events (AES) and serious adverse events (SAEs) during treatment as assessed by the National Cancer Institute Standard for Common Terminology for Adverse Events (CTCAE) version 5.0 and their association with the investigational drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Yihebali Chi, Study Chair — National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital

IPD SHARING:
Plan to Share IPD: No